CLINICAL TRIAL: NCT06291454
Title: CCL19/MIP3beta and CCL20/MIP3alpha Levels in the Gingival Crevicular Fluid of the Patients With Stage III Grade B and C Periodontitis
Brief Title: GCF Levels of Chemokines in Periodontitis
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Prof.Dr. Figen ÖNGÖZ DEDE, Clinical Professor, Ordu University
Other Study IDs: 741100
Record Dates: First submitted 2024-02-22; First posted 2024-03-04 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stage III Grade B periodontitis group (Group 1): Stage III Grade B periodontitis patients and systemically healthy
  Interventions: Diagnostic Test: Routine periodontal examination
- Stage III Grade C periodontitis group (Group 2): Stage III Grade C periodontitis patients and systemically healthy
  Interventions: Diagnostic Test: Routine periodontal examination
- Control group (Group 3): Periodontally healthy (control group) and systemically healthy patients
  Interventions: Diagnostic Test: Routine periodontal examination

INTERVENTIONS:
Diagnostic Test: Routine periodontal examination — In all of the patients, the following indexes were used routinely for the periodontal examination: Sillness-Löe's plaque index (PI) (Silness & Löe, 1964), Löe-Sillness's gingival index (GI)(Löe & Silness, 1963), probing depth (PD) to measure the extent and severity of periodontal disease, clinical attachment level (CAL), and bleeding on probing (BOP)(Ainamo & Bay, 1975) to determine activity. In addition, routine radiographic evaluations were performed to determine bone levels.GCF samples were collected using standardized filter papers.

SUMMARY:
This study aimed to determine CCL19/MIP3beta(β) and CCL20/MIP3alpha(α) in the gingival crevicular fluid (GCF) of the patients with different periodontitis phenotypes.

A total of 72 individuals, 24 with Stage III Grade B periodontitis (Group 1), 24 with Stage III Grade C periodontitis (Group 2), and 24 periodontally healthy (control group) (Group 3), were included in the study. GCF and clinical periodontal parameters were obtained at baseline. MIP3β and MIP3α levels in GCF were determined by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 20 natural teeth, excluding third molars.
* Periodontitis patients had at least two non-adjacent sites per quadrant with probing depth (PD) ≥ 5 mm and clinical attachment level (CAL) ≥ 5 mm with gingival inflammation, and alveolar bone loss affecting >30% of the teeth, as detected on clinical and radiographical examinations.
* Periodontally healthy control group had no sign of gingival inflammation, no PD > 3mm and no evidence of attachment or bone loss

Exclusion Criteria:

* History of systemic disease.
* Regular use of any drugs which can effect the immune system or inflammatory response in the 6 months preceding the start of the study.
* Periodontal treatment during last 6 months that could affect periodontal status.
* Smoking.
* History of radiotherapy or chemotherapy.
* Current pregnancy, lactation or menopause.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Group 1: Stage III Grade B periodontitis group
  * Group 2: Stage III Grade C periodontitis group
  * Group 3: Periodontally healthy control group
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
CCL19/MIP3beta(β) levels | Baseline
  CCL19/MIP3beta(β) levels in the gingival crevicular fluid (GCF) of the all groups
CCL20/MIP3alpha(α) levels | Baseline
  CCL20/MIP3alpha(α) levels in the gingival crevicular fluid (GCF)

SECONDARY OUTCOMES:
CCL19/MIP3beta(β) levels and clinical parameters | Baseline
  Correlation between CCL19/MIP3beta(β) levels in the gingival crevicular fluid (GCF) of the all groups and all clinical parameters
CCL20/MIP3alpha(α) levels and clinical parameters | Baseline
  Correlation between CCL20/MIP3alpha(α) levels in the gingival crevicular fluid (GCF) of the all groups and all clinical parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Faculty of Dentistry, Ordu, Turkey (Türkiye)